CLINICAL TRIAL: NCT03250156
Title: Investigating Train the Trainer Delivery of Mindfulness-based Training- Ft. Drum Soldiers
Brief Title: Investigating Train the Trainer Delivery of Mindfulness-based Training
Acronym: TTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Fort Drum (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amishi Jha, Associate Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20120450
Record Dates: First submitted 2017-07-25; First posted 2017-08-15 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Resilience; Stress
Keywords: Mindfulness; Attention; Working Memory; Psychological Well-Being; Proctored Practice
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We aim to recruit three groups. Two groups will receive mindfulness training (MBAT) but will differ in their level of duty day support to engage in daily assigned mindfulness exercises. The Proctored group (n = 45) will receive mindfulness training and complete assigned exercises during the duty day, integrated into their daily physical training. The Non-Proctored group (n = 45) will receive identical mindfulness training, but complete their assigned exercises on their own time. These participants will not receive additional duty day support for their practice. A third group will receive no training and serve as a control group (No-Training Control, n = 45).
  The design relies on group randomization at the level of individual platoons. This is due to the military requirement that organic unit structure is maintained during testing and course session scheduling. The number of participants is based on prior research (Jha et al., 2017).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBAT with proctored practice (Experimental): Participants will engage in Mindfulness Based Attention Training (MBAT) in 4, 2-hour training classes with 1 class per week. Participants in the proctored practice group will complete assigned, out of class mindfulness exercises during the duty day - for example, as part of their daily physical training (e.g., mindful cooldown, final 15 minutes of PT is spent engaging in a mindfulness exercise using a guided recording).
  Interventions: Behavioral: MBAT with proctored practice
- MBAT with non-proctored practice (Active Comparator): Participants will engage in Mindfulness Based Attention Training (MBAT) in 4, 2-hour training classes with 1 class per week. Participants in the non-proctored practice group will complete assigned, out of class mindfulness exercises on their own time with no structured duty day support.
  Interventions: Behavioral: MBAT with non-proctored practice
- No Training Control (No Intervention): This group will receive no intervention.

INTERVENTIONS:
Behavioral: MBAT with proctored practice — The training program is known as Mindfulness-Based Attention Training, or MBAT. The MBAT program is based on the principles of Mindfulness-Based Stress Reduction, but contextualized for military personnel using themes relevant to military life. The training content is comprised four central themes: concentration, body awareness, open monitoring, and compassion. Participants will have proctored practice and complete the assigned, out-of-class mindfulness exercises during the duty day as party of their physical training.
  Arms: MBAT with proctored practice
Behavioral: MBAT with non-proctored practice — The training program is known as Mindfulness-Based Attention Training, or MBAT. The MBAT program is based on the principles of Mindfulness-Based Stress Reduction, but contextualized for military personnel using themes relevant to military life. The training content is comprised four central themes: concentration, body awareness, open monitoring, and compassion.Participants will not have proctored practice and will complete the assigned, out-of-class mindfulness exercises on their own.
  Arms: MBAT with non-proctored practice

SUMMARY:
This project aims to evaluate the effectiveness of mindfulness training (MT) on cognitive and psychological factors when incorporated to the duty-day schedule of servicemembers (via proctored mindfulness practice). Based on prior literature, it can be hypothesized that the benefits of MT on measures of attention, working memory, and psychological well-being will be greater for servicemembers who engage in proctored mindfulness practice and receive duty-day support compared to servicemembers who practice independently, on their own time, with no structured duty day support.

DETAILED DESCRIPTION:
Background: Prior research on mindfulness training (MT) in military servicemembers showed that MT can effectively protect against degradation in attention and working memory over high-demand intervals. The benefits of MT in servicemembers were also linked to greater engagement in mindfulness practice. These prior MT programs delivered their training via a direct delivery approach, which involved a mindfulness training expert (TE) providing training to an end-user (e.g., military servicemembers). While successful, these programs are poorly suited for rapid, large-scale dissemination because these programs require direct training from a mindfulness training expert to an end-user and a considerable amount of time dedicated to training. To overcome these issues, the principal investigator together with a mindfulness expert developed a mindfulness training program contextualized for the U.S. Army, known as MBAT (Mindfulness-Based Attention Training), that is amenable to the train-the-train delivery approach and can provide rapid, large-scale dissemination to thousands of individuals. Specifically, Master Resilience Trainer - Performance Expert specialists (PEs), who have extensive experience working with soldiers but no mindfulness experience, were trained to deliver the MBAT course.

Problem: While training PEs to deliver MBAT complies with the U.S. Army time constraints, it remains unclear what is the best way to incorporate daily mindfulness practice into the duty schedule of servicemembers, which has a pivotal contribution to the protection against decline over high-demand intervals.

Project Goal: The aim of the present study is to investigate the impact of proctored vs. non-proctored practice of MBAT delivered by a PE to servicemembers. To investigate this issue, a trained PE will deliver MBAT to two groups of soldiers who will differ in the amount of duty-day support received to complete out-of-class mindfulness exercises. One group will be assigned proctored practice incorporated in the daily physical training (PT) and another group will be assigned non-proctored practice during which participants will perform the exercise independently, on their own.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Active duty military
* Able to understand and provide signed informed consent

Exclusion Criteria:

* Non-controlled severe medical disease that might interfere with the performance of the study.
* Any other condition the investigator might deem problematic for the inclusion of the volunteer in a trial of this nature will also be considered.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Change in Sustained Attention to Response Task (SART) | Participants will complete the SART at three time points: Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  The SART is used to assess attentional performance and self-reported mind wandering (i.e., off-task thinking which is typically self-generated and compromises the performance of the task at hand). The task uses a continuous performance paradigm involving button presses to frequently presented non-targets (numbers 1, 2, 4, 5, 6, 7, 8, and 9) but requires the participants to withhold their response to the infrequent target (number 3). Withholding responses only to infrequent targets encourages a pre-potent response and mind wandering. Real-time subjective experience of mind wandering during SART is assessed through experience-sampling probes randomly presented throughout the task.
Change in Working Memory Task with Affective Distraction (WMDA) | Participants will complete the WMDA at three time points: Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  The WMDA is used to assess the ability to hold information in working memory while overcoming emotional reactivity and distraction. Specifically, participants are presented with a memory item that they need to memorize and hold in memory during a delay interval. During the delay, emotionally negative or neutral scene images are presented. The negative images are combat scenes from Iraq or Afghanistan (Morey et al., 2009) and the neutral images are non-combat scenes.

SECONDARY OUTCOMES:
Change in Positive and Negative Affect Scale (PANAS) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  PANAS assesses positive and negative affect. It consists of a list of descriptors of positive (e.g., 'interested', 'enthusiastic') and negative (e.g., 'irritable', 'upset') affects. Items are rated on a 5-point scale (1 = very slightly or not at all, 5 = extremely), according to how participants feel. The Positive Affect scale reflects the extent to which a person feels enthusiastic, active, and alert; the Negative Affect scale reflects unpleasant mood states, such as anger, disgust, and fear.
Change in Perceived Stress Scale (PSS) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  PSS assesses the degree to which situations in one's life are viewed as stressful within the past month. Individual items assess feelings of stress, nervousness, irritation at life's hassles, and perceptions of one's own coping and control over a situation.

OTHER OUTCOMES:
Change in Connor-Davidson Resilience Score (CD-RISC) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  CD-RISC assesses an individual's tendency to cope with change and pressure in a productive way.
Change in Five-Facet Mindfulness Questionnaire (5FMQ) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  5FMQ assesses five major measures of mindfulness, including non-judgment of experience, non-reactivity to inner experience, observing emotions, acting with awareness, and describing feelings in words.
Change in Combat Experiences Scale (CES) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  CES assesses combat experiences in the military context.
Change in PTSD Checklist_Military (PCLM) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  PCLM assesses the symptoms of Post-Traumatic Stress Disorder in military personnel
Change in The Pittsburgh Sleep Quality Index (PSQI) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  A self-rated questionnaire which assesses sleep quality and disturbances in seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual PSQI assesses sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Change in Interpersonal Reactivity Index (IRI) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  The empathic concern subscale of the IRI is a 7-item measure used to gauge feelings of empathy towards others.
Change in Self-Compassion Scale (SCQ) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  A 26-item measure used to measure aspects of self-compassion.
Change in Obsessive Compulsion Index (OCI-R) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  An 18-item scale used to assess symptoms of Obsessive-Compulsive Disorder.
Change in Center for Epidemiological Studies Depression Scale (CES-D) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  This 20-item scale measures the major components of depressive symptomatology in the general population (i.e., nonpsychiatric persons older than 18).
Change in Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) | Pre-intervention baseline (T1), post-intervention up to 2 weeks after the end of the 4-week training (T2), and follow-up up to two months after the end of the training (T3).
  An alcohol screen that identifies people who are hazardous drinkers or have active alcohol use disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Amishi P Jha, Ph.D, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Coral Gables, Florida
  - Ft. Drum, Fort Drum, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jha, AP, Morrison, AB, Parker, SC, & Stanley, EA. Practice is protective: Mindfulness training promotes cognitive resilience in high-stress cohorts. Mindfulness. 2016; 7(1), 1-13. doi: 10.1007/s12671-015-0465-9.
- [Background] Jha AP, Morrison AB, Dainer-Best J, Parker S, Rostrup N, Stanley EA. Minds "at attention": mindfulness training curbs attentional lapses in military cohorts. PLoS One. 2015 Feb 11;10(2):e0116889. doi: 10.1371/journal.pone.0116889. eCollection 2015. PMID 25671579
- [Background] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Background] Jha AP, Witkin JE, Morrison AB, Rostrup N, Stanley E. Short-Form Mindfulness Training Protects Against Working Memory Degradation over High-Demand Intervals. Journal of Cognitive Enhancement 2017 1(2): 154-171. doi:10.1007/s41465-017-0035-2.